CLINICAL TRIAL: NCT01935154
Title: Phase II Study of Vx001 Vaccine in HLA-A*0201 Positive Patients With TERT Positive Stage IV or Recurrent Stage I-III NSCLC
Brief Title: Efficacy Study of Vx001 Vaccine in NSCLC Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vaxon Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Vx-001-201
Record Dates: First submitted 2013-08-26; First posted 2013-09-04 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Non-small Cell Lung Cancer Metastatic
Keywords: NSCLC; Vaccine
MeSH Terms: interventions — telomerase reverse transcriptase p572Y, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo will be administered evey 3 weeks from w0 to W15 than every 12 weeks until disease progression.
  Interventions: Drug: Placebo
- Vx-001 (Experimental): Vx-001 will be administered evey 3 weeks from w0 to W15 than every 12 weeks until disease progression.
  Interventions: Drug: Vx-001

INTERVENTIONS:
Drug: Vx-001
  Arms: Vx-001
Drug: Placebo
  Arms: Placebo

SUMMARY:
Patients with stage IV or recurrent stage I-III NSCLC with documented disease control (objective response or stable disease) within 3 weeks after platinum based 1st line chemotherapy; only HLA-A*0201 positive patients with TERT expressing tumors will be included.

The objective of the trial is survival rate at 12 months.

ELIGIBILITY:
Main Inclusion Criteria:

1. Male or female ≥18 years of age;
2. Documented stage IV NSCLC as defined by IASLC Lung Cancer Staging Project (7th edition) or recurrent stage I-III disease at least 6 months after resection or after the end of adjuvant chemotherapy or after standard locoregional treatment as defined by the American College of Chest Physicians;
3. Patients treated with 4 cycles platinum based 1st line chemotherapy as defined by the American College of Chest Physicians (i.e. radiotherapy are not allowed except palliative radiotherapy of bone metastasis);
4. Documented HLA-A*0201 positivity, as determined by a local laboratory;
5. TERT-positive NSCLC, as assessed by a central laboratory; for this, availability of adequate tissue biopsy from the primary tumor, lymph nodes or distant metastases is a prerequisite;
6. CR, PR, or SD according to RECIST 1.1 criteria after the completion of platinum-based first-line chemotherapy;
7. ECOG performance status 0, 1;

Main Exclusion Criteria:

1. Mixed small cell and NSCLC histologies;
2. Patients with stage IV or recurrent NSCLC who have been previously treated with therapy other than platinum-based first-line chemotherapy;
3. Prior treatment with cancer vaccines;
4. Prior treatment with immunotherapy (e.g., interferons, interleukins, TNF, or biological response modifiers, such as GM-CSF etc) within four weeks prior to randomization;
5. Prior treatment with hormone (including corticosteroids) within 2 weeks prior to randomization;
6. Prior treatment with any investigational drugs, within 4 weeks prior to randomization;
7. Patients with brain metastases;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2012-08; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Time-to-event comparison of overall survival (OS) in Vx-001 treated vs placebo treated patients. | 12 months

SECONDARY OUTCOMES:
Overall survival rate | 12 months
Comparison of Time to Treatment Failure in Vx-001 treated vs placebo treated patients. | Traitement failure

OTHER OUTCOMES:
Comparison of vaccine induced immune responses between Vx-001 vs placebo in terms of frequency of TERT specific IFN-γ and perforin producing T cells in the blood of patients. | week 18

CONTACTS AND LOCATIONS:
Overall Officials: Vassilis Georgoulias, MD,PhD, Principal Investigator — Iaso General Hospital
Locations (70):
- Czechia (2):
  - Fakultni nemocnice Plzen, Plzen-Bory
  - Vseobecna fakultni nemocnice, Prague
- France (5):
  - University Hospital of Angers, Angers
  - Ambroise Paré Hospital, Boulogne-Billancourt
  - Hopital Nord, Marseille
  - Pitié-Salpetrière Hospital, Paris
  - Pontchaillou Hospital, Rennes
- Germany (10):
  - Hospital Grosshansdorf, Großhansdorf
  - Lungenklinik Hemer, Hemer
  - Klinikum Kassel GmbH, Kassel
  - University Medical center Kiel, Kiel
  - Klinik Löwenstein, Löwenstein
  - Chirurgische Klinik-Inderdisziplinäre Thorakale Oncologie, Mannheim
  - Mühlenkreiskliniken (AöR) Johannes Wesling Klinikum Minden, Minden
  - LMU Klinikum der Universität München, Munich
  - Pius Hospital Oldenburg, Oldenburg
  - Mathias Spital Rheine Medizinische Klinik V, Rheine
- Greece (12):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - 251 General Airforce Hospital, Athens
  - General hospital of thoracic diseases Sotiria, Athens
  - Aretaieio Hospital, Athens
  - General Hospital Alexandra, Athens
  - Iaso General Hospital Cholargos, Athens
  - University Hospital of Heraklion, Heraklion
  - University General Hospital of Ioannina, Ioannina
  - General Oncology Hospital of Kifissia Agioi Anargyroi, Nea Kifissia
  - University Hospital of Patras, Rio
  - University General Hospital Papageorgiou, Thessaloniki
  - General Hospital G. Papanikolaou, Thessaloniki
- Italy (11):
  - SG Moscati Hospital, Avellino
  - G. Rummo Hospital, Benevento
  - Mater Domini Catanzaro Hospital, Catanzaro
  - European Institute of Oncology, Milan
  - San Paolo Hospital, Milan
  - Seconda Universita degli Studi Napoli Hospital, Naples
  - Insituto Oncologico Veneto, Padua
  - S. Maria della Misericordia Hospital, Perugia
  - A.O.U di Pisa Hospital, Pisa
  - S. Maria Nuova Hospital, Reggio Emilia
  - University Hospital of Siena, Siena
- Poland (11):
  - Uniwersytet Medyczny Bialistok, Bialystok
  - Hospicjum im. ks. T. Dutkiewicza SAC, Gdansk
  - Przychodnia KOMED, Konin
  - Nzoz Vesalius, Krakow
  - MS Clinsearch, Lublin
  - Oddział Onkologii z Pododdziałem Chemioterapii Nowotworów Płuc, Olsztyn
  - Mazowieckie Centrum Leczenia Chorób Płuc i Gruźlicy w Otwocku, Otwock
  - Med-Polonia, Poznan
  - Specjalistyczny Szpital im. prof.Alfreda Sokołowskiego, Szczecin
  - Centrum Onkologii - Instytut im. M. Skłodowskiej - Curie, Warsaw
  - Fundacja Hospicjum Onkologiczne św. Krzysztofa, Warsaw
- Romania (9):
  - SC Oncopremium Team SRL, Baia Mare
  - Spit. Jud. de Urgenţă, Brăila
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Institutului Oncologic "Prof. Dr. I. Chiricuţă" Cluj-Napoca, Cluj-Napoca
  - Medisprof SRL, Cluj-Napoca
  - Oncolab SRL, Craiova
  - Spitalul Clinic Judetean de Urgenta Sibiu, Sibiu
  - Spitalul Clinic Judetean de Urgenta "Sf. Ioan cel Nou", Suceava
  - Oncomed SRL, Department of Medical Oncology, Timișoara
- Spain (10):
  - USP Institut Universitari Dexeus, Barcelona
  - University Hospital P. Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu I Sant Pau, Barcelona
  - Ico-Hospital Germans Trias I Pujol, Barcelona
  - Hospital Provencial de Castellón, Castellon
  - Oncologia Medica FUNDACIÓN JIMÉNEZ DÍAZ, Madrid
  - Hospital Univesitario Puerta de Hierro, Madrid
  - H.R.U. Carlos Haya Málaga, Málaga
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Clinico de Valencia, Valencia

REFERENCES:
- [Derived] Gridelli C, Ciuleanu T, Domine M, Szczesna A, Bover I, Cobo M, Kentepozidis N, Zarogoulidis K, Kalofonos C, Kazarnowisz A, Korozan M, de Las Penas R, Majem M, Chella A, Griesinger F, Bournakis E, Sadjadian P, Kotsakis A, Chinet T, Syrigos KN, Correale P, Gallou C, Jamet JM, Vetsika EK, Kosmatopoulos K, Georgoulias V; Vx-001-201 trial team. Clinical activity of a htert (vx-001) cancer vaccine as post-chemotherapy maintenance immunotherapy in patients with stage IV non-small cell lung cancer: final results of a randomised phase 2 clinical trial. Br J Cancer. 2020 May;122(10):1461-1466. doi: 10.1038/s41416-020-0785-y. Epub 2020 Mar 25. PMID 32210365